CLINICAL TRIAL: NCT00862550
Title: Randomized Pilot Trial of Acupuncture for Prevention of Radiation-Induced Xerostomia
Brief Title: Xerostomia Pilot Fudan: Acupuncture for Prevention of Radiation-Induced Xerostomia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-0801; NCI-2009-01558 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Head and Neck Cancer; Xerostomia
Keywords: Head and Neck Cancer; HNC; Nasopharyngeal carcinoma; Acupuncture; Radiation-Induced Xerostomia; Xerostomia; Dry Mouth; Radiation
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia; Nasopharyngeal Carcinoma | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Acupuncture (Areas known to help dry mouth)
  Interventions: Other: Acupuncture
- Group 2 (Experimental): Acupuncture (Areas not known to help dry mouth)
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — 20 Minute Acupuncture Sessions Before Radiation Therapy Treatment, 3 Days Per Week for 7 Weeks.

SUMMARY:
PRIMARY AIM

1. Determine the feasibility of providing true and sham acupuncture treatment to patients at Fudan University Cancer Hospital (Cancer Hospital) who are receiving radiation treatment for cancer of the head and/or neck area.

   SECONDARY AIMS
2. Determine if true acupuncture is more effective than sham acupuncture for preventing radiation-induced xerostomia among cancer patients at Cancer Hospital.
3. Determine if true acupuncture is more effective than sham acupuncture for reducing the severity of radiation-induced xerostomia.

DETAILED DESCRIPTION:
Acupuncture is the use of very thin needles that are stuck in your skin at certain areas of the body, acupuncture is believed to affect bodily function.

Screening Tests:

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will have a physical exam.
* You will complete 3 short questionnaires about your quality-of-life and current saliva flow. It will take about 5 minutes to complete all the questionnaires.
* Two (2) saliva samples will be collected. To collect the first saliva sample, you will collect saliva in a vial (small tube or jar) for 5 minutes, by allowing saliva to collect in your mouth and then spitting it into the vial. You will wait 5 minutes and then hold a sour liquid in your mouth for 1 minute. Then a second saliva sample will be collected.
* A traditional Chinese medicine diagnosis will be performed. During this diagnosis, your pulse will be checked and photographs of your tongue will be taken. You will not be able to be identified by the photos. The photos will be destroyed when the study is complete. This will allow a more objective check of your tongue condition.
* Women who are able to become pregnant must have a negative urine pregnancy test.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

Study Groups:

If you are found to be eligible to take part in the study, you will be randomly assigned (as in the flip of a coin) into 1 of 2 groups. Both groups will have acupuncture sessions for 20 minutes before radiation therapy treatments.

* If you are in Group 1, you will have the needles stuck in areas that are known to help dry mouth.
* If you are in Group 2, you will have the needles stuck in areas that are not known to help dry mouth.

When the study is over, participants in Group 2 will be offered 1 week of acupuncture (3 treatments) in the areas known to help dry mouth.

Acupuncture:

All acupuncture sessions will be done before your radiation therapy 3 days a week for 7 weeks. The acupuncturist will put in the needles in certain areas of your body (including your chin, wrist, leg, and ear) while you are lying on a bed. The needles will remain in your body for about 20 minutes.

Study Visits:

Both groups will have the following tests and procedures performed before each acupuncture treatment, once a week:

* Your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be measured.
* You will be asked about any drugs you may be taking.
* You will complete the same questionnaires that you filled out during the screening tests.

Saliva samples will be collected on Weeks 1, 3, 4, 6, and 7. The samples will be collected the same way as done in screening. The samples will be collected after the acupuncture sessions on Weeks 1, 4, and before the acupuncture on Weeks 3 and 6.

You will have the Chinese medicine diagnosis on Weeks 3 and 7.

Length of Study:

You will be on study for 11 weeks. You will be taken off study if the condition gets worse or if intolerable side effects occur. You will be taken off study if you take any drugs for dry mouth.

End-of-Study Visit:

You will have an end-of-study visit 1 month after your last radiation treatment (Week 11). The following tests and procedures will be performed:

* Your vital signs will be measured.
* You will be asked about any drugs you may be taking.
* You will complete the quality-of-life and saliva flow questionnaires.
* You will have the 2 saliva samples a saliva sample will be collected.
* You will have the Chinese medicine diagnosis.

This is an investigational study. Up to 23 patients will take part in this study. All will be enrolled at the Fudan University Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:1) Adult >/= 18 year of age and able to sign informed consent

2) Diagnosed with nasopharyngeal carcinoma and scheduled to undergo IMRT

3) Treatment plan must include treatment at a mean dose of 25 gray or more bilateral to the parotid

4) Must have anatomically intact parotid and submandibular glands

5) Karnofsky Performance Status > 60

6) If the participant is female and of child bearing potential, must have a negative urine pregnancy test. (Acupuncture should be used cautiously during pregnancy since some points have been shown to stimulate uterine contractions

Exclusion Criteria:

1. History of xerostomia prior to the head and neck radiation therapy (Sjögren's disease or other underlying systemic illness known to cause xerostomia).
2. Prior head and neck radiation treatment
3. Suspected or confirmed physical closure of salivary gland ducts on either side
4. Known bleeding disorders or on Heparin or Coumadin
5. Upper or lower extremity deformities that could interfere with accurate acupoint location or alter the energy pathway as defined by traditional acupuncture theory
6. Local skin infections at or near the acupuncture site or active systemic infection
7. History of cerebrovascular accident or spinal cord injury. (The mechanism of action for acupuncture may be associated with central nervous system (CNS) activity, and patients with CNS pathology may respond differently to treatment than the general population.)
8. Mental incapacitation or significant emotional or psychiatric disorder that, in the opinion of the investigator, precludes study entry as these patients may not be able to cooperate with this slightly invasive procedure or with the data collection process
9. Current acknowledged use of any illicit drugs or evidence of alcohol abuse as defined by The American Psychiatric Association criteria
10. Participants who are taking or who have taken any investigational new drug within the last 30 days, or who are planning to take such a drug during the course of the study
11. Current acknowledged use of other alternative medicines such as herbal preparations that could affect salivary function. Each patient will be asked for a list of herbal supplements they are currently taking and this will be reviewed on an individual basis. Patients will be excluded if they are taking any herbs known or suspected to affect salivary function
12. Participants taking amifostine, cholinergic agonist medication (Pilocarpine, Cevimeline), beta adrenergic antagonists, anticholinergic agents, saliva substitutes or other medications known to affect salivary function
13. Currently receiving acupuncture for any condition
14. Prior use of acupuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2009-03 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Subject Recruitment (#) | 2 Years
  Feasibility determined by how many eligible patients approached consented to be in the trial and patients' reported satisfaction with the study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S. Chiang, MD, MS, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org